CLINICAL TRIAL: NCT00460746
Title: Open Label Phase 3b, 48 wk Pilot Study of the Antiviral Efficacy and Tolerability of Combination of PREZISTA/r and TMC125 When Substituted for Enfuvirtide, Current Protease Inhibitor(s) and NNRTI(s) in Antiretroviral Resistant Patients With Viral Suppression But Who Are Intolerant of Enfuvirtide.
Brief Title: Enfuvirtide/Current Protease Inhibitor Switch to PREZISTA (Darunavir)/Ritonavir + TMC125 in HIV Patients With Enfuvirtide Side Effects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011866; TMC114HIV3009 (Other: Tibotec, Inc.)
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: HIV
Keywords: HIV; AIDS; Immunodeficiency Virus, Human; PREZISTA; darunavir; TMC114; TMC125; Protease Inhibitor; Non-Nucleoside Reverse Transcriptase Inhibitor; enfuvirtide; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): TMC125, Darunavir; RitonavirTMC125-200mg two times a day for 48 weeks; Darunavir -200mg two times a day for 48 weeks; Ritonavir-100mg two times a day for 48 weeks;
  Interventions: Drug: TMC125, Darunavir; Ritonavir

INTERVENTIONS:
Drug: TMC125, Darunavir; Ritonavir — TMC125-200mg two times a day for 48 weeks; Darunavir -200mg two times a day for 48 weeks; Ritonavir-100mg two times a day for 48 weeks;

SUMMARY:
The purpose of this study is to examine the safety, tolerability, and effectiveness of darunavir/ritonavir combined with TMC125 when current protease inhibitor(s), Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI(s)) and enfuvirtide are replaced by darunavir/ritonavir and TMC125 in HIV positive patients who can no longer tolerate enfuvirtide and are experiencing viral suppression. Other antiviral drugs in the regimen are to remain unchanged.

DETAILED DESCRIPTION:
This is a multi-center, open-label (doctors and patients know which drug is being given), Phase IIIb clinical trial to evaluate the effectiveness, safety and tolerability of the combination of PREZISTA (darunavir)/ritonavir and TMC125 when substituted for enfuvirtide, current protease inhibitor(s) and Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI(s)) in antiretroviral resistant patients with viral suppression but who are intolerant of enfuvirtide. This study will be conducted in the U.S. at up to 5 sites where 40 patients will receive PREZISTA (darunavir) /ritonavir twice daily (600/100mg) and TMC125 (200 mg) twice daily over a 48-week treatment period.

The study will consist of a total of 11 patient visits. At the screening visit (Week -1 to -6) blood will be collected from patients to determine eligibility. Once all data are available to determine the eligibility of the patient, the baseline visit will be scheduled and trial treatment initiated at this visit. The Baseline Visit (Day 1) will be followed by a 48-week treatment period. The patient will be evaluated at Weeks 2, 4, 8, 12, 16, 24, 36, and 48. Patients will be asked to return for a 2-week follow up visit at Week 50.

Treatment will include PREZISTA (darunavir) /ritonavir and TMC125 plus continued nucleosides. The patient must continue all existing nucleosides in their background regimen for the duration of the study.

During the treatment period, the patient will be seen at regular visits during which the investigator will assess the patient's medical condition, any Adverse Events and study drug compliance. Laboratory evaluations for efficacy and safety will be done at regular visits. Study patients will receive oral (by mouth) PREZISTA (darunavir) 600 mg and 100 mg of ritonavir twice a day in combination with TMC125 200mg orally twice a day for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 positive
* History of drug resistance or antiretroviral failure while receiving each of three drug classes: Nucleoside Reverse Transcriptase Inhibitors (NRTIs), Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) and (protease inhibitors) PIs
* On a PI containing regimen with enfuvirtide with HIV viral load (VL) < 400 copies/mL for 6 months or longer
* Continuously using the same PI regimen for 4 months prior to Screening
* Decline to continue enfuvirtide or their physician recommends discontinuation due to injection site reactions that persist despite optimal technique and training with available methods of administration or loss of sites for injection due to tissue nodules and hardening.

Exclusion Criteria:

* No use of any drug contraindicated in the current US package insert for PREZISTA (darunavir) or in the investigators brochure for TMC125
* No prior or current therapy with PREZISTA (darunavir) or TMC125
* No prior genotypic results demonstrating 3 or more darunavir resistance-associated mutations associated with diminished response to darunavir (V11I, V32I, L33F, I47V, I50V, I54L, I54M, G73S, L76V, I84V or L89V). Patients with > 3 darunavir resistance-associated mutations with available darunavir phenotypes, may be enrolled if the resistance phenotype demonstrates: Fold Change (FC) <10 to darunavir by PhenoSense GT (Monogram Biosciences) or FC <10 to darunavir by Antivirogram (Virco, BVBA) or FC <3.4 to darunavir by vircoTYPE (Virco BVBA)
* AST or ALT >5 times ULN
* Calculated CrCl < 30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc
Locations (1):
- Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Darunavir(TMC114)/Eravirine(TMC125): Darunavir/ritonavir (DRV/r) combined with Etravirine ([ETR] also known as TMC125) when current protease inhibitor(s) (PIs), non-nucleoside reverse transriptase inhibitor(s) (NNRTIs), and enfuviritide (ENF) were replaced by DRV/r and ETR in subjects with intolerance to ENF.
Period: Overall Study
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Started | 10
Completed | 8
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
Age Continuous [Median (Full Range); unit: years] | 48 [35 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6
  Hispanic | 4
Viral Load <50 copies/mL [Number; unit: participants] | 10
CD4 count [Median (Full Range); unit: cells/mm^3] | 301 [187 to 663]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Maintain Plasma HIV Viral Load Measurements < 400 Copies/ml at 2, 4, 8, 12, 16, 24, 36 and 48 Weeks After Switching to DRV/r and ETR, Missing Equals Failure.
Time Frame: 48 weeks
Population: ITT population. One subject (001) who discontinued due to adverse events had a VL < 50 copies/mL at Week 4. Another subject (013) who was lost to follow-up had VL <50 copies/mL through Week 36.
Measure: Number; unit: percentage of participants
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
percentage of participants
  Baseline (Day 1) | 100
  Week 2 | 100
  Week 4 | 100
  Week 8 | 90
  Week 12 | 80
  Week 16 | 90
  Week 24 | 90
  Week 36 | 90
  Week 48 | 80
  Post-Treatment Follow Up | 90

2. Secondary Outcome: Proportion of Patients Who Have Viral Load Measurements <50 Copies/ml at 2, 4, 8, 12, 16, 24, 36 and 48 Weeks After Switching to DRV/r and ETR, Missing Equals Failure.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
percentage of participants
  Baseline (Day 1) | 100
  Week 2 | 90
  Week 4 | 90
  Week 8 | 90
  Week 12 | 80
  Week 16 | 90
  Week 24 | 90
  Week 36 | 90
  Week 48 | 80
  Post-Treatment Follow Up | 90

3. Secondary Outcome: CD4+ Cell Count (x 10^6 Cell/L): Baseline and Median Changes From Baseline at 4, 8, 12, 16, 24, 36 and 48 Weeks.
Time Frame: Week 48
Population: Intent To Treat (ITT), last observation carried forward (LOCF).
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
cells/mm^3
  Baseline (Day 1) | 301.0 [187.0 to 663.0]
  Week 4 Change from Baseline | -12.0 [-32.0 to 61.0]
  Week 8 Change from Baseline | -32.0 [-169.0 to 81.0]
  Week 12 Change from Baseline | -17.0 [-100.0 to 61.0]
  Week 16 Change from Baseline | -7.0 [-73.0 to 81.0]
  Week 24 Change from Baseline | 19.0 [-36.0 to 71.0]
  Week 36 Change from Baseline | 38.0 [-59.0 to 117.0]
  Week 48 Change from Baseline | 63.5 [-53.0 to 100.0]

4. Secondary Outcome: CD4+ Cell Count (x 10^6 Cell/L): Baseline and Mean Changes From Baseline at 4, 8, 12, 16, 24,36 and 48 Weeks.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
cells/mm^3
  Baseline (Day 1) | 338.3 (135.91)
  Week 4 Change from Baseline | 2.3 (31.22)
  Week 8 Change from Baseline | -25.0 (72.04)
  Week 12 Change from Baseline | -18.9 (44.25)
  Week 16 Change from Baseline | 0.5 (53.58)
  Week 24 Change from Baseline | 24.5 (34.00)
  Week 36 Change from Baseline | 22.7 (58.84)
  Week 48 Change from Baseline | 47.3 (48.03)

5. Secondary Outcome: Median Change From Baseline in Triglycerides at Week 48.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
mg/dL
  Baseline (Day 1) | 229.0 [121.0 to 402.0]
  Week 48 Change from Baseline | -24.5 [-227.0 to 78.0]

6. Secondary Outcome: Median Change From Baseline in Total Cholesterol at Week 48.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
mg/dL
  Baseline (Day 1) | 189.0 [159.0 to 244.0]
  Week 48 Change from Baseline | -27.5 [-44.0 to 27.0]

7. Secondary Outcome: Median Change From Baseline in LDL Cholesterol at Week 48.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
mg/dL
  Baseline (Day 1) | 100.0 [63.0 to 149.0]
  Week 48 Change from Baseline | -9.0 [-30.0 to 17.0]

8. Secondary Outcome: Median Change From Baseline in HDL Cholesterol.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
mg/dL
  Baseline (Day 1) | 47.5 [25.0 to 54.0]
  Week 48 Change from Baseline | -2.5 [-15.0 to 10.0]

9. Secondary Outcome: Median Change From Baseline in Total Cholesterol (TC) / High Denisty Lipoprotein (HDL) Ratio at Week 48.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: ratio of TC and HDL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
ratio of TC and HDL
  Baseline (Day 1) | 4.7 [2.94 to 6.40]
  Week 48 Change from Baseline | -0.3 [-0.82 to 1.20]

10. Secondary Outcome: Median Change From Baseline in Glucose at Week 48.
Time Frame: Week 48
Population: ITT , LOCF.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Number analyzed (Participants) | 10
mg/dL
  Baseline (Day 1) | 92.5 [74.0 to 105.0]
  Week 48 Change from Baseline | 1.0 [-21.0 to 12.0]

ADVERSE EVENTS:
Arm/Group | Darunavir(TMC114)/Eravirine(TMC125)
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darunavir(TMC114)/Eravirine(TMC125) (N=10)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) — Noted by investigator as doubtfully related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darunavir(TMC114)/Eravirine(TMC125) (N=10)
Abdominal pain upper (General disorders) | 1 (1) — Relationship is other than not related.
Amnesia (Nervous system disorders) | 1 (1) — Relationship is other than not related.
Constipation (Gastrointestinal disorders) | 1 (1) — Relationship is other than not related.
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) — Relationship is other than not related.
Depression (Psychiatric disorders) | 2 (2) — Relationship is other than not related.
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Relationship is other than not related.
Diarrhea (Gastrointestinal disorders) | 3 (3) — Relationship is other than not related.
Disturbance in attention (Nervous system disorders) | 1 (1) — Relationship is other than not related.
Diverticulitis (Infections and infestations) | 1 (1) — Relationship is other than not related.
Dizziness (Nervous system disorders) | 1 (1) — Relationship is other than not related.
Dry mouth (Gastrointestinal disorders) | 1 (1) — Relationship is other than not related.
Fatigue (General disorders) | 4 (4) — Relationship is other than not related.
Headache (Nervous system disorders) | 3 (3) — Relationship is other than not related.
Heart rate increase (Vascular disorders) | 1 (1) — Relationship is other than not related.
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) — Relationship is other than not related.
Hypertension (Vascular disorders) | 2 (2) — Relationship is other than not related.
Insomnia (Psychiatric disorders) | 2 (2) — Relationship is other than not related.
Nausea (Gastrointestinal disorders) | 1 (1) — Relationship is other than not related.
Pain (General disorders) | 1 (1) — Relationship is other than not related.
Rash (Skin and subcutaneous tissue disorders) | 3 (3) — Relationship is other than not related.
Somnolence (Nervous system disorders) | 1 (1) — Relationship is other than not related.

LIMITATIONS AND CAVEATS:
Conclusions on efficacy and safety are limited as the target enrollment of 40 subjects was not reached due to a shortage of eligible subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If TTCA does not publish within 12 months after study conclusion or after TTCA confirms there will be no multicenter publication, Institution may publish their results from their site individually, provided TTCA has 60 day review for confidentiality and additional 60 day delay for patent application.